CLINICAL TRIAL: NCT01426204
Title: Efficacy, Safety and Adherence of Patients Infected With Hepatitis C Virus in Retreat With INFERGEN (Interferon Alfacon1)
Acronym: OBSERVER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Closter Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: COL-BIO-NIS001
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Retreatment; Failures; Infergen; Interferon Alfacon-1
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a Phase 4, descriptive, observational, open, prospective study of patients who their doctor prescribes INFERGEN for clinical practice. No medication was provided by the sponsor. The planned observation time is 48 weeks and 24 weeks of follow-up.

Each investigator participating in this registry will employ his or her discretion and standard clinical practice to determine when to see the patient in the clinic, how to manage the patient's drug regimen, and how best to monitor the patient's response and tolerance to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to consent to data being collected
2. Considered by the investigator as an appropriate patient for treatment with INFERGEN in retreatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Gastrointestinal Practices as well as hepatologyst practice. Academic Centers have been asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of SVR | 24 weeks post end of therapy
  •Determine the incidence of SVR, defined as undetectable HCV RNA measured 24 weeks after therapy ends, associated with prescribed, therapy with Infergen® (Interferon alfacon 1) in patients chronically infected with HCV, in retreatment.

SECONDARY OUTCOMES:
Safety profile | Treatment weeks 4, 12, 24,32, 40, 48, and Follow-Up weeks 4 and 24
  •Capture of defined adverse events (AEs),dose changes or cessation, and adherence to the prescribed dose of Infergen and other prescribed therapies over the course of treatment